CLINICAL TRIAL: NCT04633005
Title: Polypill Strategy for the Evidence-Based Management of Heart Failure With Reduced Ejection Fraction in an Underserved Patient Population
Brief Title: Polypill Strategy for Heart Failure With Reduced Ejection Fraction
Acronym: POLY-HF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ambarish Pandey, Assistant Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTexasSouthwestern
Record Dates: First submitted 2020-11-02; First posted 2020-11-17 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure
Keywords: heart failure; adherence; LVEF; GDMT
MeSH Terms: conditions — Heart Failure | interventions — Tin Fluorides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Polypill Arm (Experimental): Participants will be randomized to receiving a fixed-dose polypill in addition to other guideline-directed medical therapies prescribed by their physician. Polypill formulations will include metoprolol succinate (a beta-blocker), empagliflozin (an SGLT2-inhibitor), and spironolactone (a mineralocorticoid antagonist). Four dose formulations of the pill, varied in metoprolol succinate dose (25, 50, 100, 150 mg), will be available for up-titration of the beta-blocker dose per ACC/AHA/HFSA guidelines.
  Interventions: Drug: Polypill
- Usual Care (Active Comparator): Participants in the usual care arm received individual components of GDMT with initiation and up-titration performed in partnership with their primary outpatient physician teams
  Interventions: Drug: Control Rx

INTERVENTIONS:
Drug: Polypill — Polypill formulation consisting of metoprolol succinate, empagliflozin, and spironolactone.
  Arms: Polypill Arm
Drug: Control Rx — Typical prescriptions of guideline-directed therapies for heart failure with reduced ejection fraction.
  Arms: Usual Care

SUMMARY:
Heart failure with a reduced ejection fraction (HFrEF) represents a significant public health burden in the United States, with a growing prevalence particularly among African Americans and Hispanic Americans and individuals of low socioeconomic status (SES). Although effective therapies exist, gaps in their uptake contribute substantially to the excess burden of heart failure. The "polypill" is an inexpensive once daily pill containing three agents proven to improve morbidity and mortality in heart failure and represents potential strategy for increasing the utilization of proven HF therapies. The proposed study is a pragmatic, single-center, randomized trial to test the feasibility and effectiveness of a polypill-based strategy for the treatment of HFrEF in a low-income, racially diverse population.

DETAILED DESCRIPTION:
Heart failure poses a major public health challenge in the United States. It affects more than 6.2 million people and is the leading cause of hospitalization among older adults, with a growing prevalence among Black, Hispanic, and low-income populations.

Despite advances in the treatment of heart failure, the associated morbidity and mortality remain high. From the time of heart failure diagnosis, survival is approximately 50% at 5-years and 10% at 10-years.8 Improved mortality and hospitalization rates have been observed due to the advent of mortality-reducing HFrEF therapies and earlier diagnosis. Nonetheless, substantial gaps in the uptake of guideline-directed medical therapies (GDMT) exist. GDMT, which include beta-blockers (BB), angiotensin converting enzyme inhibitors (ACEI), angiotensin receptor blockers (ARB), and mineralocorticoid receptor antagonists (MRA), have been demonstrated to reduce all-cause mortality by > 50% when used in combination. Nonetheless, fewer than 25% of eligible patients currently receive these medications at any dose, with socially disadvantaged groups having the lowest rates of utilization.

The polypill is an alternative management strategy. The polypill combines multiple evidence-based medications in a single pill, which reduces pill burden and improves adherence. Therapy with multiple medications can be conveniently initiated at an early stage of disease, increasing the overall therapeutic benefit accrued over time. This is particularly relevant in settings where patients experience barriers to care due to high cost burden with copays associated with medication initiation, frequent lab tests, and need for multiple follow up visits.

Polypills have been shown to be feasible and effective in multiple settings, including in the prevention and treatment of cardiovascular disease (CVD). They have been well tolerated and additionally demonstrate significant improvements in adherence when compared to usual therapies in randomized control trials. However, no randomized trial to date has evaluated a polypill strategy for the treatment of heart failure, a condition in which pill burden and adherence pose substantial challenges to management.

The proposed study is a single-center, randomized trial to test the feasibility and effectiveness of a polypill-based strategy for the treatment of HFrEF (EF ≤40%) in a low-income population. The setting for our proposed study is Parkland Hospital in Dallas, Texas, a large county hospital that serves a racially diverse, uninsured population. We will utilize 4 distinct polypill formulations to allow for up-titration of the beta-blocker component of the polypill. The pill will contain spironolactone 12.5 mg, empagliflozin 10 mg, and 25 mg, 50 mg, 100 mg, or 150 mg of metoprolol succinate. The once-daily polypill will be added to baseline therapy with a renin-angiotensin system antagonist (ACEI, ARB, or ARNI).

We hypothesize that use of a polypill-based strategy in HFrEF will be feasible and lead to improved left ventricular systolic function compared with usual care. These hypotheses will be tested in the following aims:

Primary Aim: To determine whether the use of a polypill for HFrEF leads to higher left ventricular ejection fraction (LVEF) compared with usual care in a low-income population. The primary endpoint will be the change in LVEF, obtained by cardiac MRI (CMR), from baseline to 6 months. CMR provides the greatest accuracy and reproducibility of the non-invasive cardiac imaging modalities.

Secondary Aim: To determine whether the use of a polypill for HFrEF leads to lower circulating NT-proBNP levels compared with usual care in a low-income population. Changes in circulating NT-proBNP concentrations from baseline to 6-months will be compared in participants randomized to the polypill vs usual care arm.

The primary endpoint is the change in LVEF over 6 months, based on prior studies demonstrating measurable changes in systolic function and cardiac biomarkers with treatment with GDMT. LVEF will be assessed using cardiac MRI at baseline and the end of the study period. We hypothesize that polypill use will be associated with greater improvement in LVEF compared with usual care. Secondary endpoints include a hierarchical, composite, win-ratio based endpoint consisting of: all-cause mortality, ≥5 point change KCCQ-OSS, HF hospitalization (total number), >5% change in LVEF by cardiac MRI, and having detectable levels of metoprolol succinate and/or spironolactone based on serum drug monitoring. Change in NT-proBNP, a serum marker of neurohormonal stress, is a biomarker-based secondary endpoint and a well-validated surrogate endpoint for HF trials. NT-proBNP levels have been associated with short- and long-term clinical outcomes for all stages of HFrEF and receive a class I, Level of Evidence A recommendation for diagnosis and assessment of prognosis in clinical HF guidelines. Additional secondary endpoints of interest include adherence to GDMT, as assessed by therapeutic drug monitoring and MMAS-8 score, quality of life assessed using the Kansas City Cardiomyopathy (KCCQ) Questionnaire-12, 6-minute walk distance (6-MWD), and change in LVEF assessed via echocardiogram.

The trial will be led by study investigators from the University of Texas Southwestern with joint appointments within the Parkland Health and Hospital System. The proposal builds on the team's prior experience conducting clinical trials of cardiovascular therapies in low-income, diverse populations. The trial can be performed efficiently and cost-effectively within the Parkland Health and Hospital System.

After securing permission from the clinical director and providers within the Parkland Health and Hospital System and Parkland Cardiology Clinic, the study team will begin active screening for patients with heart failure within the Parkland Cardiology Clinic and inpatient Parkland Cardiology service. We will enroll adults age ≥18 years with de novo or chronic HFrEF (LVEF ≤ 40%) with recent hospitalization or outpatient visit at Parkland who are not on target GDMT. De novo HFrEF will be defined as new-onset HFrEF with hospitalization for HF or outpatient diagnosis with 180 days of screening. Chronic HFrEF will include patients with a known diagnosis of HFrEF for more than 6 months.

To achieve the target enrollment, the study team will enroll participants during inpatient hospitalization and from outpatient clinics. Patients will be started on the polypill prior to discharge or at the first outpatient visit after heart failure hospitalization. In both settings, the polypill will be substituted for the individual component medications, with other medications continued as prescribed. The team will include a study coordinator with extensive experience performing clinical trials at Parkland Health & Hospital Systems. The team will perform pre-screening using EHR data after obtaining permission from the Parkland inpatient and clinic heart failure attendings. Patients deemed eligible for participation will be contacted prior to discharge from their HF hospitalization or at the time of their initial visit to cardiology clinic following discharge. Patients will be informed about the study, its goals, and the risks and benefits of participating, and will be invited to participate. Potential participants will be asked to fill out a questionnaire seeking information on medication use, health status, and on the characteristics to assess potential eligibility. Eligible participants may also be identified based on review of the EHR post-discharge and will be contacted through an introductory letter and pre-screening questionnaire. . Based on our initial experience, we estimate that we will need to contact 700 patients over the 4-year enrollment period to enroll 175 patients in the study. In our prior polypill trial, conducted in an outpatient setting, we observed a 45% response rate to the initial invitation, of which ~50% met eligibility criteria and consented to randomization. We will record all contact attempts and responses to determine recruitment rates and reasons for entry or non-entry into the trial. The study team has substantial experience with recruitment of participants for clinical trials and observational studies at Parkland Hospital.

Participants who meet eligibility criteria will be invited to enroll in the trial. Participants will be randomly assigned in a 1:1 ratio using a computerized algorithm. Block randomization will be performed according to baseline use of a polypill component and race/ethnicity group. The randomization key will be maintained by a faculty member with no involvement in the trial.

The study investigators will prescribe the polypill to those in the active arm. In response to the initial polypill prescription, participants will receive an initial presription containing a 30-day supply of medication. Subsequent refills of 30-day supply will be made available. Participants will be instructed to take one pill per day for the duration of the study. All polypill medication, including unopened or partially used containers, will be maintained at the study site. As this is an open-label trial, there will be no placebo provided in the usual care arm. Participants in the usual care arm will be eligible for reimbursement for co-payments for GDMT to minimize cost differentials between study arms.

In accordance with local regulatory requirements, the investigator or designated research staff will document the quantity of polypill dispensed and/or administered to study participants, the amount returned by study participants, and the amount received from and returned to the vendor when applicable. Product accountability records will be maintained throughout the course of the study. Concomitant medications and non-drug therapies not specifically prohibited by the study are allowed. All concomitant medications taken during the study will be recorded by study staff. Prohibited medications include all medications that interact with the components of the polypill or are contraindicated in patients with HFrEF.

At the baseline visit informed consent will be obtained. Responses to the baseline questionnaire will be reviewed by a study coordinator as a final check on inclusion and exclusion criteria and current medication use. A medical and social history will be obtained. Vital signs will be measured in seated participants, according to standardized protocols. A 15 mL blood sample will be obtained for eligibility laboratories. Pre-menopausal women will undergo a rapid urine pregnancy test.

At 1, 3, and 6 months post-randomization, participants will be scheduled for a follow-up visit at the outpatient clinic. At these follow-up visits, the study coordinators will review questionnaires for completeness, assess vital signs, collect a blood sample, assess medication adherence by the MMAS-8 questionnaire, assess for medication safety, tolerance, and side effects. The up-titration in GDMT or polypill beta-blocker dose will be performed, as tolerated on each visit. A 6-minute walk test and quality of life assessment using the KCCQ will be performed at each study visit. A metabolic panel test will be performed at each follow-up to assess for hyperkalemia or kidney dysfunction. Therapeutic drug monitoring of metoprolol and spironolactone will be assessed at 6 months. Additional clinic visits will be allowed at the discretion of the patients' physicians.

Subjects will receive $50 per study visit. In addition, subjects will also receive $50 for their CMR visits at baseline and follow up. Participants will also receive travel vouchers and/or transportation reimbursements for their follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Adults age > = 18 years
* HF with left ventricular ejection fraction <= 40% within 3 months of screening who are not on target dose guideline directed medical therapy
* New York Heart Association class II, III, or IV symptoms

Exclusion Criteria:

* Age < 18
* Systolic blood pressure < 110 mm Hg at enrollment if not on HTN therapy.
* Systolic blood pressure <100 mm Hg at enrollment if on HTN therapy
* Serum creatinine >2.5 for men and 2.0 for women
* Serum potassium > 5.0 mEq/L
* Current need for inotropes
* Cardiac index < 2.2 L/min/m2
* History of revascularization within 30 days or plan for revascularization
* History of type 1 diabetes mellitus
* History of allergic reaction or contraindication to a beta-blocker (BB), mineralocorticoid receptor antagonist (MRA), or sodium glucose cotransporter 2 inhibitor (SGLT2i)
* Contraindication to receive any of the components of the polypill
* Pregnancy
* < 6 month expected survival
* Inability to provide written informed consent
* Persistent or permanent atrial fibrillation who may not have optimal MRI imaging
* Extreme obesity (BMI > 45 kg/m2)
* ICD/Pacemaker devices that are incompatible with MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | 6 months
  Measured by cardiac MR

SECONDARY OUTCOMES:
Hierarchical Composite Endpoint | baseline through 6 months
  1. Hierarchical composite endpoint of all-cause mortality, ≥5 point change Kansas City Cardiomyopathy Questionnaire - Overall Summary Score (KCCQ-OSS), HF hospitalization or emergency department visit for HF (total number), >5% change in LVEF by cardiac MRI, and having detectable levels of metoprolol succinate and/or spironolactone based on therapeutic drug monitoring.
Kansas City Cardiomyopathy Questionnaire Quality of Life | Baseline, 1 month, 3 months, 6 months
  12-item Kansas City Cardiomyopathy Questionnaire measures patients' quality of life. Possible score range from 0 to 100, with higher scores indicating a better quality of life.
Medication adherence | 6-months
  Therapeutic drug monitoring of metoprolol and spironolactone.
Six-minute walk distance | baseline, 1 month, 3 months, 6 months
  Six-minute walk test
LVEF through echocardiography | 6 months
  assessed by echocardiogram
NT-ProBNP level | baseline, 1 month, 3 months, 6 months
  Serum level
Medication Adherence | This score ranges from 0-8, with 0 indicating lowest adherence and 8 indicating highest adherence. This will be assessed at baseline, 1 month, 3 month, and 6 month.
  Self-report via the Morisky Medication Adherence Score - 8
HF Events | Through 6 month follow-up
  Composite of HF hospitalization or emergency department visits for HF
Composite HF events or mortality | Through 6 month follow-up
  Composite of HF hospitalization or emergency department visits for HF or all-cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States